CLINICAL TRIAL: NCT07378410
Title: Outcomes of Intra-Operative Aspiration Vs Non-Aspiration for Distended Gallbladder in Laparoscopic Cholecystectomy
Brief Title: Role of Intra-Operative Aspiration in Distended GB in LC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aswan University (Other)
Responsible Party: Principal Investigator, Ali Hussein Abdelaal, Master degree candidate and Resident of General Surgery, Aswan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Asw.Uni./978/9/24
Record Dates: First submitted 2026-01-20; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Acute Calculous Cholecystitis; Gallbladder Empyema; Gallbladder Mucocele
Keywords: Acute Calculous Cholecystitis; Gallbladder Empyema; Gallbladder Mucocele; Distended gallbladder; Intra-operative aspiration
MeSH Terms: conditions — Cholecystitis, Acute; Cholecystitis

STUDY DESIGN:
Intervention Model Description: comparing the efficacy of intra-operative Gallbladder content aspiration in overdistended cases with completion of the operation without aspiration
Who Masked: Participant
Masking Description: Participants agreed to participate in the study and undergo the LC
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aspiration group (Experimental)
  Interventions: Procedure: Laparoscopic needle
- Non-Aspiration group (No Intervention)

INTERVENTIONS:
Procedure: Laparoscopic needle — During classic LC, either with preoperative or accidently intra-operative overdistended GB using a laparoscopic needle to decompress the GB and make the operation much easier
  Arms: Aspiration group

SUMMARY:
Laparoscopic cholecystectomy (LC) is a standard procedure for gallstones and the standard surgical approach for acute calcular cholecystitis, superseding open cholecystectomy for gallbladder (GB) pathologies. Despite this progress, mortality rates in high-risk cohorts remain substantial, ranging between 3.7% and 41.0%. Moreover, the recommended modality for mucocele which is defined as distension and marked dilatation of the GB associated with dysfunction is LC.

The routine aspiration showed significant less percentage of GB perforation during surgery with similarity for other factors . However, routine aspiration of the GB during uncomplicated LC is considered an unnecessary intervention and therefore not recommended as a routine practice.

Accidental GB perforation occurs in about 20% of laparoscopic cholecystectomies, and bile contamination in the abdominal cavity can cause SSI and lead to the formation of a residual abscess or wound infection.

Grasping a thick and distended GB is one of the most common technical difficulties of laparoscopic cholecystectomy in acute cholecystitis. If the GB is distended it should be decompressed it to avoid conversion to open due to bile duct injury or perforation with spillage of bile and gallstones previously, authors had advocated conversion if iatrogenic perforation occurred.

DETAILED DESCRIPTION:
This study was conducted on patients with symptomatic calcular cholecystitis presented to Aswan university hospital.

The following parameters were measured intraoperative difficulty.

* Operative time
* Incidence of biliary tree injury
* Higher surgeon consultation
* Conversion into open surgery All groups were followed up for 30 days period for post-operative complication clinically and by sonar.
* Wound infection
* Liver bed bleeding
* Collection in the liver bed
* Peritonitis
* Hospital stays.

ELIGIBILITY:
Inclusion Criteria:

* Patient with calcular cholecystitis, GB mucocele or GB empyema
* Distended gallbladder: shiny, over distended, long, difficult to grasp and manipulate gallbladder.
* Acute or chronic calcular cholecystitis

Exclusion Criteria:

* Obstructive jaundice
* Non distended gallbladder
* Previous upper abdomen operations
* Pregnant

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2026-01-01 (Actual); Study Completion 2026-01-01 (Actual)

PRIMARY OUTCOMES:
Difficulty of the operation | 30 days
  the difficulty will be assessed by the following Operative time, Incidence of biliary tree injury, Higher surgeon consultation and Conversion to open chole

SECONDARY OUTCOMES:
Liver bed bleeding | 30 days
  checking post procedures and postoperative through the drain
30-day mortality | 30 days
  follow-up the patient in the outpatient and by phone
Hospital stays. | 30 days
  total stay in the hospital
Peritonitis | 30 days
  incidence of peritonitis in the first week of the operation

CONTACTS AND LOCATIONS:
Overall Officials: Ali H Abdelaal, Principal Investigator — Faculty of Medicine, Aswan University
Locations (1):
- Aswan University, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barrat, C., Champault, A., Matthyssens, L., & Champault, G. (2004). L'effraction de la vésicule lors des cholécystectomies laparoscopiques n'influence pas la morbidité. Étude prospective. Annales de Chirurgie, 129(1), 25-29. https://doi.org/10.1016/j.anchir.2003.11.011
- [Background] Calik, A., Topaloglu, S., Topcu, S., Turkyilmaz, S., Kucuktulu, U., & Piskin, B. (2007). Routine intraoperative aspiration of gallbladder during laparoscopic cholecystectomy. Surgical Endoscopy and Other Interventional Techniques, 21(9), 1578-1581. https://doi.org/10.1007/s00464-006-9159-7 Guzmán-Valdivia, G. (2008). Routine Administration of Antibiotics to Patients Suffering Accidental Gallbladder Perforation During Laparoscopic Cholecystectomy is not Necessary. Surgical Laparoscopy, Endoscopy & Percutaneous Techniques, 18(6), 547-550. https://doi.org/10.1097/SLE.0b013e3181809e72 Lee, K.-T., Shan, Y.-S., Wang, S.-T., & Lin, P.-W. (2005). Verres needle decompression of distended gallbladder to facilitate laparoscopic cholecystectomy in acute cholecystitis: A prospective study. Hepato-Gastroenterology, 52(65), 1388-1392. Lisotti, A., Linguerri, R., Bacchilega, I., Cominardi, A., Marocchi, G., & Fusaroli, P. (2022). EUS-guided gallbladder drainage in high-risk surgical patients with acute cholecystitis-Procedure outcomes and evaluation of mortality predictors. Surgical Endoscopy, 36(1), 569-578. https://doi.org/10.1007/s00464-021-08318-z Majumder, A., Altieri, M. S., & Brunt, L. M. (2020). How do I do it: Laparoscopic cholecystectomy. Annals of Laparoscopic and Endoscopic Surgery, 5, 15-15. https://doi.org/10.21037/ales.2020.02.06 Mishra, R. K. (2022, June 12). Cholecystectomy for Mucocele of Gallbladder. https://www.laparoscopyhospital.com/streamvideo/index.php?pid=536&p=28 Ponsky, J. L. (1991). Complications of laparoscopic cholecystectomy. The American Journal of Surgery, 161(3), 393-395. https://doi.org/10.1016/0002-9610(91)90605-D Shea, J. A., Berlin, J. A., Bachwich, D. R., Staroscik, R. N., Malet, P. F., McGuckin, M., Schwartz, J. S., & Escarce, J. J. (1998). Indications for and Outcomes of Cholecystectomy. Annals of Surgery, 227(3), 343-350. https://doi.org/10.1097/00000658-199803000-00005 Shirah, B. H., Shirah, H. A., & Albeladi, K. B. (2018). The value of intraoperative percutaneous aspiration of the mucocele of the gallbladder for safe laparoscopic management. Updates in Surgery, 70(4), 495-502. https://doi.org/10.1007/s13304-018-0565-x Siddiqui, M. R. S., Sajid, M. S., Nisar, A., Ali, H., Zaborszky, A., & Hasan, F. (2011). A meta-analysis of outcomes after routine aspiration of the gallbladder during cholecystectomy. International Surgery, 96(1), 21-27. https://doi.org/10.9738/1361.1 Usuba, T., Nyumura, Y., Takano, Y., Iino, T., & Hanyu, N. (2017). Clinical outcomes of laparoscopic cholecystectomy with accidental gallbladder perforation. Asian Journal of Endoscopic Surgery, 10(2), 162-165. https://doi.org/10.1111/ases.12348 Wood, S., Lewis, W., & Egan, R. (2019). Optimising Surgical Technique in Laparoscopic Cholecystectomy: A Review of Intraoperative Interventions. Journal of Gastrointestinal Surgery, 23(9), 1925-1932. https://doi.org/10.1007/s11605-019-04296-9